CLINICAL TRIAL: NCT04134039
Title: A Randomized, Assessor-masked, 2-way Cross-over, Multi-centre, Clinical Investigation to Evaluate the Performance Rate of a Polyurethane Condom in Healthy Monogamous Couples When Compared With a Standard Latex Condom
Brief Title: A Clinical Investigation to Assess the Performance of a Polyurethane Condom Versus a Latex Condom in Healthy Monogamous Couples
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1003201
Record Dates: First submitted 2019-10-11; First posted 2019-10-21 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Control of Pregnancy; Prevention of Sexually Transmitted Infections
MeSH Terms: interventions — Condoms

STUDY DESIGN:
Intervention Model Description: The condom types will be tested in a 2-way cross-over design where couples will be randomised to use each of the 2 condom types in a defined order, according to the randomisation schedule.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Each condom will be individually wrapped in its primary packet then be put in an identical box. All branding will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyurethane (PU) condom (Experimental): Following randomisation each couple will be given one set of 7 condoms as per randomisation schedule. After use of at least 5 condoms, couples will return to the clinic site for collection of their next set of condoms. Each couple will test a maximum of 14 condoms during their participation in the investigation.
  Interventions: Device: Polyurethane (PU) condom; Device: Natural Rubber Latex (NRL) condom
- Natural Rubber Latex (NRL) condom (Experimental): Following randomisation each couple will be given one set of 7 condoms as per randomisation schedule. After use of at least 5 condoms, couples will return to the clinic site for collection of their next set of condoms. Each couple will test a maximum of 14 condoms during their participation in the investigation.
  Interventions: Device: Polyurethane (PU) condom; Device: Natural Rubber Latex (NRL) condom

INTERVENTIONS:
Device: Polyurethane (PU) condom — A minimum of 5 condoms (maximum 7 condoms) of each condom type will be provided to couples to be used during vaginal intercourse over a 4 week period, the assessment period. Couples will repeat the assessment period each of the 2 condom types.
Device: Natural Rubber Latex (NRL) condom — A minimum of 5 condoms (maximum 7 condoms) of each condom type will be provided to couples to be used during vaginal intercourse over a 4 week period, the assessment period. Couples will repeat the assessment period each of the 2 condom types.

SUMMARY:
This investigation is designed to evaluate the performance rate of a polyurethane (PU) condom versus a standard natural rubber latex (NRL) condom.

DETAILED DESCRIPTION:
In this clinical investigation, a new PU male condom (test condom) will be evaluated against a marketed NRL male condom (reference condom). This clinical investigation will also evaluate the in-use tolerance of the test and reference condoms.

ELIGIBILITY:
Main Inclusion Criteria:

1. A male and a female subject aged: 18 - 60 years inclusive.
2. All subjects must be generally healthy and in a mutually monogamous heterosexual relationship - current relationship ≥ 3 months.
3. All couples must be sexually active and agree to have penile-vaginal intercourse with a frequency sufficient to meet protocol requirements (a minimum of 5 coital acts over 4 weeks).
4. The female partner should already be on an established highly effective form of non-barrier contraception, unless post-menopausal.
5. Couples must agree not to use drugs or non-investigational devices that can affect sexual performance.

Main Exclusion Criteria:

1. Either partner is or becomes aware of an allergy or sensitivity to the ingredients of the test products, including the test or reference condoms.
2. Either partner has a pre-existing skin condition (severe eczema/ psoriasis) or systemic allergic reactions or as confirmed by the subject and physical examination.
3. Either partner that needs to use condoms for a specific sexually transmitted infection (STI) protection e.g. discordance for Human Immunodeficiency Virus (HIV) or herpes.
4. Subjects that have previous or planned genital surgery, that in the opinion of the Investigator would consider the subject unsuitable to participate in the clinical investigation e.g. laser for abnormal smear.
5. Male partners that have known erectile or ejaculatory dysfunction.
6. A female partner that has been diagnosed with or treated for vaginal complaints (including vaginal dryness) in the previous 3 months which, in the opinion of the investigator, deems the partner unsuitable for the investigation.
7. Any subject who has clinical symptoms or signs of a sexually transmitted diseases (STD) or HIV/ AIDS or has a previous history of high-risk behaviour as judged by the investigator.
8. Female partner using medication which in the investigator's opinion would affect vaginal mucosal secretion, such as Chlorpheniramine at any time in the 14 days (or 5 half-lives of the drug, whichever is longer) before first condom use.
9. A male partner with abnormal penile anatomy that would, in the opinion of the investigator, affect the ability to keep the condom in place during intercourse.
10. Either partner intends to continue to use antihistamines, anti-inflammatory drugs or pain killers for the duration of the investigation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 470 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Compared clinical failure rate of condom use between the test condom group and the reference condom group | within 2 hours following each coital act for each condom use
  Clinical failure rate is calculated as the number of condoms with at least 1 acute clinical failure event divided by the number of condoms used during intercourse, reported as a percentage. Clinical failure events, defined in ISO 29943-1:2017, will be reported by subjects.

SECONDARY OUTCOMES:
Performance (clinical slippage rate) of the Polyurethane (PU) condom | within 2 hours following each coital act for each condom use
  Clinical slippage rate is calculated as the number of condoms with at least 1 clinical slippage event divided by the number of condoms used during intercourse, reported as a percentage. Clinical slippage events, defined in ISO 29943-1:2017, will be reported by subjects.
  A clinical slippage is defined as a condom slipping off completely during intercourse or during withdrawal from the vagina. Slippage that occur because the user failed to hold onto the condom at the base of the penis during withdrawal and/ or because the user delayed withdrawal after sex are to be record as "non-clinical slippage", these events are considered user failures.
Performance (clinical slippage rate) of the Natural Rubber Latex (NRL) condom | within 2 hours following each coital act for each condom use
  Clinical slippage rate is calculated as the number of condoms with at least 1 clinical slippage event divided by the number of condoms used during intercourse, reported as a percentage. Clinical slippage events, defined in ISO 29943-1:2017, will be reported by subjects.
  A clinical slippage is defined as a condom slipping off completely during intercourse or during withdrawal from the vagina. Slippage that occur because the user failed to hold onto the condom at the base of the penis during withdrawal and/ or because the user delayed withdrawal after sex are to be record as "non-clinical slippage", these events are considered user failures.
Performance (clinical breakage rate) of the Polyurethane (PU) condom | within 2 hours following each coital act for each condom use
  Clinical failure rate is calculated as the number of condoms with at least 1 acute clinical failure event (clinical slippage or clinical breakage) divided by the number of condoms used during intercourse, reported as a percentage. Clinical failure events, defined in ISO 29943-1:2017, will be reported by subjects.
Performance (clinical breakage rate) of the Natural Rubber Latex (NRL) condom | within 2 hours following each coital act for each condom use
  Clinical failure rate is calculated as the number of condoms with at least 1 acute clinical failure event (clinical slippage or clinical breakage) divided by the number of condoms used during intercourse, reported as a percentage. Clinical failure events, defined in ISO 29943-1:2017, will be reported by subjects.
Incidence of treatment-emergent adverse events and adverse device effects, defined in MEDDEV 2.7/3 | 12 weeks
Subject's experience on the use of each type of condoms [Acceptability and Tolerability | 12 weeks
  Acceptability and tolerability as assessed by subject perceived questionnaires (designed by following ISO 29943-1)

CONTACTS AND LOCATIONS:
Overall Officials: Unnop Jaisamrarn, MD, Principal Investigator — King Chulalongkorn Memorial Hospital
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No